CLINICAL TRIAL: NCT04793191
Title: Predicting Acute Postoperative Pain by the Preoperative Lower Back Pain in the Gynecological Laparoscopy
Brief Title: Predicting Acute Postoperative Pain by the Preoperative Lower Back Pain
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, Associate professor, The Catholic University of Korea
Other Study IDs: back pain
Record Dates: First submitted 2021-03-09; First posted 2021-03-11 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2021-03

CONDITIONS: Benign Gynecological Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate if the level of preoperative lower back pain has the effect on the acute postoperative pain after gynecological laparoscopy

ELIGIBILITY:
Inclusion Criteria:

* women scheduled for elective gynecological laparoscopy

Exclusion Criteria:

* psychiatric disease eg. anxiety, depression, etc.
* diagnosed as cancer
* the use of vasoactive drug
* chronic pain except lower back pain

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the women scheduled for elective gynecological laparoscopy in the tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
the intensity of acute postoperative pain | during 30 min in the recovery room
  The intensity of pain is assessed using the numeric rating scale (0=no pain; 10=the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Young Eun Moon, MD, PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine
Locations (1):
- Seoul St.Mary's Hospital, Seoul, Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: No